CLINICAL TRIAL: NCT02958839
Title: The Relationship Between Fibroblast Growth Factor 23 and the Recurrence of Atrial Fibrillation After Catheter Ablation: a Nested Case-Control Study
Brief Title: Relationship Between Fibroblast Growth Factor 23 and Recurrence of Atrial Fibrillation After Catheter Ablation
Acronym: REBECCA
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Zhongkai Zhao, intern of cardiology, Peking University Third Hospital
Other Study IDs: L03-ZZK-FGF23
Record Dates: First submitted 2016-11-04; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Fibroblast Growth factor 23
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be obtained by a peripheral venipuncture and will be centrifuged at 3,200 *g for 10 minutes at approximately 4℃ within an hour of collection. The serum will be separated into aliquots and stored at -80℃ until personnel blinded to the patients' clinical information performed the analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Recurrence Group: In the case control trial, patients who have any episode of atrial fibrillation/atrial flutter/atrial tachycardia after a blanking period of 3 months from the catheter ablation procedure will be assign to the recurrence group
  Interventions: Procedure: Catheter ablation
- Non-recurrence Group: In the case control trial, patients who do not have any episode of atrial fibrillation/atrial flutter/atrial tachycardia after a blanking period of 3 months from the catheter ablation procedure will be assign to the recurrence group
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Procedure: Catheter ablation — Patients with persistent or paroxysmal atrial fibrillation will go through catheter ablation

SUMMARY:
To investigate whether fibroblast growth factor 23 can be used to predict recurrence after catheter ablation for atrial fibrillation and to provide an objective basis for the clinical selection of the optimal patients for catheter ablation.

DETAILED DESCRIPTION:
Atrial fibrillation, which can result in stroke and thromboembolism in an approximately 5-fold increased risk, has been a great burden to health care system with the aging of population. Catheter ablation is the most promising treatment of atrial fibrillation. However, the recurrence rates of AF after catheter ablation are high, ranging from 20%-60%. Therefore, non-invasive predictors for AF recurrence after catheter ablation is necessary to select the optimal patients for this procedure.

Fibroblast growth factor-23 (FGF-23) is a bone-derived hormone that plays a central role in phosphate homeostasis. Recent study showed that fibroblast growth factor 23 plays an important role in cardiac remodeling and is considered to be independently associated with the occurrence of atrial fibrillation. In this study, we are going to observe the relationship between the serum FGF-23 and the arrythmia recurrence after catheter ablation of AF.

This research is going to recruit 200 consecutive patients with a history of atrial fibrillation for 180-360 days who intend to undergo catheter ablation. The day before catheter ablation, serum FGF-23 level will be detected. Echocardiogram and left atrial CT scan will also be performed on the day before catheter ablation. All patients will be routinely follow up in the outpatient department by cardiologists every month for 1 year. If patients complain about palpitations, fatigue, or other symptoms related to arrhythmia, Holter monitoring will be performed. Patients will also be advised to see their doctor anytime they have these symptoms and to undergo a 12-lead ECG examination or 24-hour Holter monitoring. In asymptomatic patients, 24-hour Holter monitoring or 7-day cardiac event recording will be performed every three months after the procedure. The endpoint for follow-up is the recurrence of atrial fibrillation, which is considered to be any episode of AF/AFL/AT after a blank period of 3 months after the procedure of catheter ablation. Those who develop recurrence of AF during follow up will be assigned to recurrence group, and those who do not develop recurrence of AF during follow up will be assigned to non-recurrence group. Comparison of the serum FGF-23 level between the two groups will be carried out in order to investigate the relationship between serum FGF-23 level and the recurrence of AF.

ELIGIBILITY:
Inclusion Criteria:

* Have a history of atrial fibrillation for 180 to 360 days
* Provide written informed consent, having understood the benefits and risks of participation in the trial

Exclusion Criteria:

* Significant structural heart disease (including symptomatic coronary heart disease; prosthetic mitral or tricuspid valve; congenital heart disease where abnormality or its correction prohibits or increases the risk of ablation)
* Atrial Fibrillation precipitated by other diseases (such as thyrotoxicosis)
* Severe dysfunction of liver or kidney
* Diabetes
* Malignant tumor
* Inability or refusal to provide written informed consent for the study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This research is going to recruit 200 consecutive patients with a history of atrial fibrillation for 180-360 days who intend to undergo catheter ablation. Atrial fibrillation is diagnosed according to guidelines; Patients with structural heart disease; renal or hepatic impairment; neoplastic disorders; atrial fibrillation precipitated by other diseases such as thyrotoxicosis; or diabetes will be excluded.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of the recurrence of atrial fibrillation | after 3 months from the procedure of catheter ablation
  The recurrence of atrial fibrillation is considered to be any episode of AF/AFL/AT after a blank period of 3 months after the procedure of catheter ablation

SECONDARY OUTCOMES:
Plasma fibroblast growth factor 23 levels | after 3 months from the procedure of catheter ablation
  Fibroblast Growth Factor 23 plays an important role in cardiac remodeling and is considered to be independently associated with the occurrence of atrial fibrillation
CHA2DS2-VASc score | after 3 months from the procedure of catheter ablation
  CHA2DS2-VASc score is used to measure the risk of thrombotic event in patient with atrial fibrillation
Cardiac CT evaluation | after 3 months from the procedure of catheter ablation
  To evaluate the degree of fibrosis of the left and right atrium and pulmonary veins

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, MD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Meng L, Yang Y, Zhang Z, Li G, Liu T. Predictive value of circulating fibroblast growth factor-23 on atrial fibrillation: A meta-analysis. Int J Cardiol. 2016 May 1;210:68-71. doi: 10.1016/j.ijcard.2016.02.100. Epub 2016 Feb 18. No abstract available. PMID 26942328